CLINICAL TRIAL: NCT00154921
Title: Clinical Usefulness of Optical Skin Biopsy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government); National Health Research Institutes, Taiwan (Other)
Other Study IDs: 9361700212; NTUH-94M29
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-11-23 (Estimated); Status verified 2004-01

CONDITIONS: Skin Neoplasms
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Traditional biopsy requires the removal, fixation, and staining of tissues from the human body. Its procedure is invasive and painful. Non-invasive in vivo optical biopsy is thus required, which should provide non-invasive, highly penetrative, three-dimensional (3D) imaging with sub-micron spatial resolution. Optical biopsy based on scanning two-photon fluorescence microscopy (TPFM) is a good method for biopsy of skin due to its high lateral resolution, low out-of-focus damage, and intrinsic three-dimensional (3D) section capability. However current technology still presents several limitations including low penetration depth, in-focus cell damages, and multi-photon phototoxicity due to high optical intensity in the 800 nm wavelength region, and toxicity if exogenous fluorescence markers were required. We study the harmonics optical biopsy of a human skin sample using a femtosecond Cr:forsterite laser centered at 1230 nm. Higher harmonics generation is known to leave no energy deposition to the interacted matters due to their energy-conservation characteristic. This energy-conservation characteristic provides the "noninvasive" nature desirable for clinical imaging. In our study, we will evaluate the clinical applications of optical skin biopsy using harmonic generation microscopy.

DETAILED DESCRIPTION:
Traditional biopsy requires the removal, fixation, and staining of tissues from the human body. Its procedure is invasive and painful. Non-invasive in vivo optical biopsy is thus required, which should provide non-invasive, highly penetrative, three-dimensional (3D) imaging with sub-micron spatial resolution. Optical biopsy based on scanning two-photon fluorescence microscopy (TPFM) is a good method for biopsy of skin due to its high lateral resolution, low out-of-focus damage, and intrinsic three-dimensional (3D) section capability. However current technology still presents several limitations including low penetration depth, in-focus cell damages, and multi-photon phototoxicity due to high optical intensity in the 800 nm wavelength region, and toxicity if exogenous fluorescence markers were required. We study the harmonics optical biopsy of a human skin sample using a femtosecond Cr:forsterite laser centered at 1230 nm. Higher harmonics generation is known to leave no energy deposition to the interacted matters due to their energy-conservation characteristic. This energy-conservation characteristic provides the "noninvasive" nature desirable for clinical imaging. In our study, we will evaluate the clinical applications of optical skin biopsy using harmonic generation microscopy.

ELIGIBILITY:
Inclusion Criteria:

* Skin lesions admitted for surgical resection.

Exclusion Criteria:

* none

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2004-01; Study Completion 2007-12

CONTACTS AND LOCATIONS:
Overall Officials: Wen-jeng Lee, M.D., Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan